CLINICAL TRIAL: NCT04466267
Title: The Molecular Mechanism of RAS Wild-type Metastatic Colorectal Cancer (mCRC) Resistance to Anti Epidermal Growth Factor Receptor (EGFR) Antibody
Brief Title: The Molecular Mechanism of RAS Wild-type mCRC Resistance to Anti-EGFR-antibody
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ruihua Xu, Clinical Professor, Sun Yat-sen University
Other Study IDs: anti-EGFR-antibody
Record Dates: First submitted 2020-07-06; First posted 2020-07-10 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tissues and peripheral blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Establishing the genetic map of primary and secondary resistance of Chinese wild RAS colorectal cancer received anti-EGFR treatment through tissues and peripheral blood NGS testing. Combination genetic data with clinical characteristics, prognosis and treatment data to explore the molecular mechanism of resistance of anti-EGFR-antibody.

DETAILED DESCRIPTION:
Cetuximab is a chimeric (mouse/human) monoclonal antibody, an epidermal growth factor receptor (EGFR) inhibitor. Many large clinical trials demonstrated that for RAS wild-type metastatic colorectal cancer (mCRC), especially left-sided RAS wild-type mCRC, cetuximab can prolong OS. But some of patients have primary resistance to cetuximab and for all patients received cetuximab will develop secondary resistance. Cell-free or circulating tumour DNA (ctDNA) including primary site and metastatic site genetic information, which can avoid tumor heterogeneity. The results of paired test detection of tissue and ctDNA showed there is 93% consistency in RAS testing. Therefore, dynamic monitoring ctDNA during anti-EGFR targeted treatment of RAS wild-type mCRC patients can implement prognosis of efficacy and response evaluation in real-time. Besides, it can monitor the variation features of resistance gene and find resistance gene in real-time. According the situation of gene change to find potential drug resistance mechanism and formulate individualization treatment plan.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years, ≤75 years, all gender;
2. Histologically proven metastatic adenocarcinoma of colorectal cancer, no previous history of cancer;
3. The clinical data of patient is intact;
4. The data of patients after surgery is intact, and the prognosis follow-up data of patient is available.

Exclusion Criteria:

1. Previous history of cancer；
2. Intact clinical data or diagnosis results of histopathology is unavailable;
3. Time of progression disease after treatment and follow-up data are unavailable;
4. Patient received blood transfusion within 3 months;
5. Other situation that researchers think it will impact the results of trails or violate ethics.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RAS wild-type metastatic colorectal cancer patients treatment with FOLFOX/FORFIRI + cetuximab
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-07-04 (Actual)

PRIMARY OUTCOMES:
The molecular mechanism of patients primary or secondary resistance to cetuximab | up to 36 months
  Dynamic monitoring ctDNA to identify potential molecular mechanism of RAS wild-type mCRC patients primary or secondary resistance to cetuximab

CONTACTS AND LOCATIONS:
Overall Officials: Ying Jin, MD.,PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Medical Oncology,Sun Yat-sen University Cancer Center, Guanzhou, Guangdong, China

REFERENCES:
- [Background] Venook AP, Niedzwiecki D, Lenz HJ, Innocenti F, Fruth B, Meyerhardt JA, Schrag D, Greene C, O'Neil BH, Atkins JN, Berry S, Polite BN, O'Reilly EM, Goldberg RM, Hochster HS, Schilsky RL, Bertagnolli MM, El-Khoueiry AB, Watson P, Benson AB 3rd, Mulkerin DL, Mayer RJ, Blanke C. Effect of First-Line Chemotherapy Combined With Cetuximab or Bevacizumab on Overall Survival in Patients With KRAS Wild-Type Advanced or Metastatic Colorectal Cancer: A Randomized Clinical Trial. JAMA. 2017 Jun 20;317(23):2392-2401. doi: 10.1001/jama.2017.7105. PMID 28632865
- [Background] Stintzing S, Modest DP, Rossius L, Lerch MM, von Weikersthal LF, Decker T, Kiani A, Vehling-Kaiser U, Al-Batran SE, Heintges T, Lerchenmuller C, Kahl C, Seipelt G, Kullmann F, Stauch M, Scheithauer W, Held S, Giessen-Jung C, Moehler M, Jagenburg A, Kirchner T, Jung A, Heinemann V; FIRE-3 investigators. FOLFIRI plus cetuximab versus FOLFIRI plus bevacizumab for metastatic colorectal cancer (FIRE-3): a post-hoc analysis of tumour dynamics in the final RAS wild-type subgroup of this randomised open-label phase 3 trial. Lancet Oncol. 2016 Oct;17(10):1426-1434. doi: 10.1016/S1470-2045(16)30269-8. Epub 2016 Aug 27. PMID 27575024
- [Background] Tejpar S, Stintzing S, Ciardiello F, Tabernero J, Van Cutsem E, Beier F, Esser R, Lenz HJ, Heinemann V. Prognostic and Predictive Relevance of Primary Tumor Location in Patients With RAS Wild-Type Metastatic Colorectal Cancer: Retrospective Analyses of the CRYSTAL and FIRE-3 Trials. JAMA Oncol. 2017 Feb 1;3(2):194-201. doi: 10.1001/jamaoncol.2016.3797. PMID 27722750
- [Background] Batth IS, Mitra A, Manier S, Ghobrial IM, Menter D, Kopetz S, Li S. Circulating tumor markers: harmonizing the yin and yang of CTCs and ctDNA for precision medicine. Ann Oncol. 2017 Mar 1;28(3):468-477. doi: 10.1093/annonc/mdw619. PMID 27998963
- [Background] Vidal J, Muinelo L, Dalmases A, Jones F, Edelstein D, Iglesias M, Orrillo M, Abalo A, Rodriguez C, Brozos E, Vidal Y, Candamio S, Vazquez F, Ruiz J, Guix M, Visa L, Sikri V, Albanell J, Bellosillo B, Lopez R, Montagut C. Plasma ctDNA RAS mutation analysis for the diagnosis and treatment monitoring of metastatic colorectal cancer patients. Ann Oncol. 2017 Jun 1;28(6):1325-1332. doi: 10.1093/annonc/mdx125. PMID 28419195